CLINICAL TRIAL: NCT00434642
Title: A Phase III, Multicenter, Randomized, Blinded, Placebo-controlled Trial of Carboplatin and Gemcitabine Plus Bevacizumab in Patients With Platinum-sensitive Recurrent Ovary, Primary Peritoneal, or Fallopian Tube Carcinoma
Brief Title: A Study of Carboplatin and Gemcitabine Plus Bevacizumab in Patients With Ovary, Peritoneal, or Fallopian Tube Carcinoma
Acronym: OCEANS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVF4095g
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Results first posted 2011-11-03 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-07

CONDITIONS: Ovarian Cancer
Keywords: Avastin; Ovarian carcinoma; Peritoneal carcinoma; Peritoneal cancer; Fallopian tube cancer; Fallopian tube carcinoma; OCEANS
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Carboplatin; Gemcitabine; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Carboplatin and gemcitabine + bevacizumab (Experimental): Carboplatin (AUC 4 mg/mL/minute) was administered intravenously (IV) on Day 1 of each of six 21-day treatment cycles. The carboplatin dose was calculated to reach a target area under the curve (AUC) of concentration x time according to the Calvert formula. Gemcitabine 1000 mg/m^2 was administered IV on Days 1 and Day 8 of each of the six 21-day treatment cycles. Bevacizumab 15 mg/kg was administered IV on Day 1 of each of the six 21-day treatment cycles. The bevacizumab dose was based on the patient's weight at baseline and remained the same throughout the study.
  Interventions: Drug: Carboplatin; Drug: Gemcitabine; Drug: Bevacizumab
- Carboplatin and gemcitabine + placebo (Active Comparator): Carboplatin (AUC 4 mg/mL/minute) was administered intravenously (IV) on Day 1 of each of six 21-day treatment cycles. The carboplatin dose was calculated to reach a target area under the curve (AUC) of concentration x time according to the Calvert formula. Gemcitabine 1000 mg/m^2 was administered IV on Days 1 and Day 8 of each of the six 21-day treatment cycles. Placebo was administered by IV on Day 1 of each of the six 21-day treatment cycles.
  Interventions: Drug: Carboplatin; Drug: Gemcitabine; Drug: Placebo

INTERVENTIONS:
Drug: Carboplatin — Carboplatin was provided as commercially available drug.
Drug: Gemcitabine — Gemcitabine was provided as commercially available drug.
Drug: Bevacizumab — Bevacizumab was supplied as a clear to slightly opalescent, sterile liquid in glass vials (400 mg in 8 mL [25 mg/mL]) with a vehicle consisting of sodium phosphate, trehalose, polysorbate 20, and Sterile Water for Injection, USP.
  Other Names: Avastin
  Arms: Carboplatin and gemcitabine + bevacizumab
Drug: Placebo — Placebo consisted of the vehicle for bevacizumab without the antibody and contained sodium phosphate, trehalose, polysorbate 20, and Sterile Water for Injection, USP.
  Arms: Carboplatin and gemcitabine + placebo

SUMMARY:
This is a placebo-controlled, randomized, multicenter Phase III study that will evaluate the safety and efficacy of bevacizumab, administered in combination with carboplatin with gemcitabine, in women with platinum-sensitive recurrent epithelial ovarian, primary peritoneal, or fallopian tube carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age ≥ 18 years
* Documented ovarian, primary peritoneal, or fallopian tube carcinoma that has recurred
* No prior chemotherapy in the recurrent setting
* Measurable disease
* Recovered from prior radiation therapy or surgery

Exclusion Criteria:

* Prior chemotherapy treatment for recurrent ovarian, primary peritoneal, or fallopian tube carcinoma
* History of abdominal fistula, gastrointestinal perforation (GIP), or intra-abdominal abscess
* Patients with clinical symptoms or signs of gastrointestinal (GI) obstruction or who require parenteral hydration, parenteral nutrition, or tube feeding
* Patients with evidence of abdominal free air not explained by paracentesis or recent surgical procedure
* Current, recent, or planned participation in an experimental drug study
* History of systemic bevacizumab (Avastin) or other vascular endothelial growth factor (VEGF) or VEGF receptor-targeted agent use
* Inadequately controlled hypertension
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association Class II or greater congestive heart failure (CHF)
* History of myocardial infarction or unstable angina
* History of stroke or transient ischemic attack (TIA)
* Known central nervous system (CNS) disease except for treated brain metastasis
* Significant vascular disease or recent peripheral arterial thrombosis
* History of hemoptysis
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2007-04; Primary Completion 2010-09 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amreen Husain, MD, Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Aghajanian C, Goff B, Nycum LR, Wang YV, Husain A, Blank SV. Final overall survival and safety analysis of OCEANS, a phase 3 trial of chemotherapy with or without bevacizumab in patients with platinum-sensitive recurrent ovarian cancer. Gynecol Oncol. 2015 Oct;139(1):10-6. doi: 10.1016/j.ygyno.2015.08.004. Epub 2015 Aug 10. PMID 26271155
- [Derived] Vaughan S, Coward JI, Bast RC Jr, Berchuck A, Berek JS, Brenton JD, Coukos G, Crum CC, Drapkin R, Etemadmoghadam D, Friedlander M, Gabra H, Kaye SB, Lord CJ, Lengyel E, Levine DA, McNeish IA, Menon U, Mills GB, Nephew KP, Oza AM, Sood AK, Stronach EA, Walczak H, Bowtell DD, Balkwill FR. Rethinking ovarian cancer: recommendations for improving outcomes. Nat Rev Cancer. 2011 Sep 23;11(10):719-25. doi: 10.1038/nrc3144. PMID 21941283

RESULTS

PARTICIPANT FLOW:
Period: Blinded Treatment Phase
Arm/Group | Carboplatin and Gemcitabine + Placebo | Carboplatin and Gemcitabine + Bevacizumab
Started | 242 | 242
Completed | 0 | 13
Not Completed | 242 | 229
Not completed — Adverse Event | 12 | 58
Not completed — Clinical Disease Progression | 4 | 5
Not completed — Disease Progression Per RECIST | 168 | 109
Not completed — Physician Decision | 19 | 27
Not completed — Sponsor's Decision To Terminate Study | 3 | 0
Not completed — Subject's Decision-Discontinue Treatment | 32 | 29
Not completed — Did not Receive Treatment | 4 | 1
Period: Open-label Treatment Phase
Arm/Group | Carboplatin and Gemcitabine + Placebo | Carboplatin and Gemcitabine + Bevacizumab
Started | 0 | 12 (One participant did not continue into the open-label treatment phase.)
Completed | 0 | 1
Not Completed | 0 | 11
Not completed — Adverse Event | 0 | 5
Not completed — Disease Progression Per RECIST | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carboplatin and Gemcitabine + Placebo | Carboplatin and Gemcitabine + Bevacizumab | Total
Number analyzed (Participants) | 242 | 242 | 484
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (10.2) | 60.5 (9.8) | 61.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 242 | 242 | 484
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) as Determined by the Investigator, Per Response Evaluation Criteria for Solid Tumors (RECIST)
Description: PFS was defined as the time from randomization to disease progression (PD), as determined by the investigator, or death due to any cause. PD: At least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started; the appearance of 1 or more new lesions; and/or the unequivocal progression of existing non-target lesions. Lesions were assessed by computed tomography (CT), magnetic resonance imaging (MRI), or ultrasound every 9 weeks.
Time Frame: From randomization through September 17, 2010 (up to 3 years, 5 months)
Population: Intent-to-treat population: All patients randomized to treatment (242 patients in each treatment group).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin and Gemcitabine + Bevacizumab | Carboplatin and Gemcitabine + Placebo
Number analyzed (Participants) | 242 | 242
Months | 12.4 [11.40 to 12.71] | 8.4 [8.31 to 9.66]
Statistical Analysis 1: Comparison: Carboplatin and Gemcitabine + Bevacizumab vs Carboplatin and Gemcitabine + Placebo; The null hypothesis was that there was no difference between the 2 treatment groups, ie, that the hazard ratio is equal to 1. The alternative hypothesis was that progression free survival was longer in the carboplatin and gemcitabine + bevacizumab group, ie, that the hazard ratio is not equal to 1; Test type: Superiority or Other; p < 0.0001, Log Rank — A P-value < 0.05 was required for significance; The analysis was stratified for time since the last platinum therapy (6-12, > 12 months) and cytoreductive surgery for recurrent disease (yes, no); Hazard Ratio (HR) = 0.484, 95% CI 2-sided [0.388 to 0.605] — The hazard ratio was estimated using Cox regression. The hazard ratio is relative to the carboplatin and gemcitabine + placebo group

2. Secondary Outcome: Percentage of Patients With an Objective Response as Determined by the Investigator, Per Response Evaluation Criteria for Solid Tumors (RECIST)
Description: An objective response was the occurrence of either a partial response (PR) or complete response (CR). PR: At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. CR: The disappearance of all target and non-target lesions. Lesions were assessed by computed tomography (CT), magnetic resonance imaging (MRI), or ultrasound every 9 weeks.
Time Frame: From randomization through September 17, 2010 (up to 3 years, 5 months)
Population: Intent-to-treat population: All patients randomized to treatment (242 patients in each treatment group).
Measure: Number; unit: Percentage of participants
Arm/Group | Carboplatin and Gemcitabine + Bevacizumab | Carboplatin and Gemcitabine + Placebo
Number analyzed (Participants) | 242 | 242
Percentage of participants | 78.5 | 57.4
Statistical Analysis 1: Comparison: Carboplatin and Gemcitabine + Bevacizumab vs Carboplatin and Gemcitabine + Placebo; The null hypothesis was that there was no difference in the percentage of patients with an objective response between the 2 treatment groups. The alternative hypothesis was that a larger percentage of patients had an objective response in the carboplatin and gemcitabine + bevacizumab group; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — A P-value < 0.05 was required for significance; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 21.1, 95% CI 2-sided [13.0 to 29.2] — The difference in response rates and the 95% confidence intervals for response rates were computed using the normal approximation to the binomial distribution

3. Secondary Outcome: Duration of Objective Response (OR) as Determined by the Investigator, Per Response Evaluation Criteria for Solid Tumors (RECIST)
Description: Duration of OR was analyzed in the subset of patients who achieved an OR. The duration of OR was defined as the time from the initial CR or PR until documented PD or death. Lesions were assessed by computed tomography (CT), magnetic resonance imaging (MRI), or ultrasound every 9 weeks.
Time Frame: From randomization through September 17, 2010 (up to 3 years, 5 months)
Population: Subset of the intent-to-treat population: All patients randomized to treatment who achieved an objective response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin and Gemcitabine + Bevacizumab | Carboplatin and Gemcitabine + Placebo
Number analyzed (Participants) | 190 | 139
Months | 10.4 [9.36 to 11.83] | 7.4 [6.31 to 8.31]

4. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization to death from any cause.
Time Frame: From randomization through July 19, 2013 (up to 6 years, 3 months)
Population: Intent-to-treat population: All patients randomized to treatment (242 patients in each treatment group).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Carboplatin and Gemcitabine + Bevacizumab | Carboplatin and Gemcitabine + Placebo
Number analyzed (Participants) | 242 | 242
Months | 33.6 [30.32 to 35.84] | 32.9 [29.80 to 37.68]
Statistical Analysis 1: Comparison: Carboplatin and Gemcitabine + Bevacizumab vs Carboplatin and Gemcitabine + Placebo; Test type: Superiority or Other; p = 0.6479, Log Rank — Summaries of duration of overall survival (median, percentiles) were estimated from Kaplan-Meier curves. The 95% confidence interval for the median was computed using the method of Brookmeyer and Crowley; The analysis was stratified for time since the last platinum therapy (≤12, >12 months) and cytoreductive surgery for recurrent disease (Yes, No); Hazard Ratio (HR) = 0.952, 95% CI 2-sided [0.771 to 1.176] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Patients Who Had a Gastrointestinal Perforation (GIP)
Description: A gastrointestinal perforation is a hole that develops through the entire wall of the stomach, small intestine, large bowel, or gallbladder.
Time Frame: From randomization through September 17, 2010 (up to 3 years, 5 months)
Population: Safety population: All patients who received at least 1 dose of protocol treatment. Due to errors in drug administration, the safety population included 247 patients in the carboplatin and gemcitabine + bevacizumab group and 233 patients in the carboplatin and gemcitabine + placebo group.
Measure: Number; unit: Percentage of participants
Arm/Group | Carboplatin and Gemcitabine + Bevacizumab | Carboplatin and Gemcitabine + Placebo
Number analyzed (Participants) | 247 | 233
Percentage of participants | 0 | 0

6. Secondary Outcome: Percentage of Patients Who Had at Least 1 Adverse Event
Time Frame: From randomization through July 19, 2013 (up to 6 years, 3 months)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Carboplatin and Gemcitabine + Bevacizumab | Carboplatin and Gemcitabine + Placebo
Number analyzed (Participants) | 247 | 233
Percentage of participants | 100.0 | 100.0

ADVERSE EVENTS:
Time Frame: From randomization through July 19, 2013
Description: Safety population: All patients who received at least 1 dose of protocol treatment. Due to errors in drug administration, the safety population included 247 patients in the carboplatin and gemcitabine + bevacizumab group and 233 patients in the carboplatin and gemcitabine + placebo group.
Arm/Group | Carboplatin and Gemcitabine + Bevacizumab | Carboplatin and Gemcitabine + Placebo
Serious Adverse Events (participants affected / at risk) | 90/247 | 59/233
Other Adverse Events (participants affected / at risk) | 246/247 | 233/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin and Gemcitabine + Bevacizumab (N=247) | Carboplatin and Gemcitabine + Placebo (N=233)
Anaemia (Blood and lymphatic system disorders) | 6 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 4
Haemolytic Uraemic Syndrome (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 3
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 8
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 2
Cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 2
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 2
Ileus Spastic (Gastrointestinal disorders) | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 3 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 4 | 6
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3
Adverse Drug Reaction (General disorders) | 1 | 1
Infusion Related Reaction (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 6
Thrombosis In Device (General disorders) | 0 | 1
Bile Duct Obstruction (Hepatobiliary disorders) | 0 | 1
Biliary Colic (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 3
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 4 | 3
Hypersensitivity (Immune system disorders) | 1 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Catheter Site Infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 2
Device Related Infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 1 | 0
Kidney Infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2
Thrombophlebitis Septic (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Viral Infection (Infections and infestations) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound Complication (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Soft Tissue Haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour Compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral Ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Haemorrhage Intracranial (Nervous system disorders) | 1 | 0
Haemorrhagic Stroke (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 1
Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 2 | 0
Speech Disorder (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 1
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Mental Status Changes (Psychiatric disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Nephrotic Syndrome (Renal and urinary disorders) | 1 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Ureteric Obstruction (Renal and urinary disorders) | 0 | 1
Female Genital Tract Fistula (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Ureteral Stent Insertion (Surgical and medical procedures) | 1 | 0
Arterial Thrombosis (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 2 | 1
Embolism (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 0
Malignant Hypertension (Vascular disorders) | 2 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombophlebitis Superficial (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 2 | 0
Vena Cava Thrombosis (Vascular disorders) | 1 | 0
Influenza Like Illness (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Embolism Venous (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin and Gemcitabine + Bevacizumab (N=247) | Carboplatin and Gemcitabine + Placebo (N=233)
Anaemia (Blood and lymphatic system disorders) | 126 | 137
Leukopenia (Blood and lymphatic system disorders) | 36 | 32
Neutropenia (Blood and lymphatic system disorders) | 172 | 158
Thrombocytopenia (Blood and lymphatic system disorders) | 135 | 111
Tinnitus (Ear and labyrinth disorders) | 14 | 11
Vision Blurred (Eye disorders) | 14 | 17
Abdominal Discomfort (Gastrointestinal disorders) | 15 | 15
Abdominal Distension (Gastrointestinal disorders) | 24 | 21
Abdominal Pain (Gastrointestinal disorders) | 60 | 58
Abdominal Pain Lower (Gastrointestinal disorders) | 20 | 16
Abdominal Pain Upper (Gastrointestinal disorders) | 19 | 17
Constipation (Gastrointestinal disorders) | 132 | 122
Diarrhoea (Gastrointestinal disorders) | 95 | 67
Dyspepsia (Gastrointestinal disorders) | 27 | 29
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 20 | 17
Gingival Bleeding (Gastrointestinal disorders) | 17 | 1
Haemorrhoids (Gastrointestinal disorders) | 18 | 6
Nausea (Gastrointestinal disorders) | 177 | 153
Rectal Haemorrhage (Gastrointestinal disorders) | 21 | 10
Stomatitis (Gastrointestinal disorders) | 39 | 16
Vomiting (Gastrointestinal disorders) | 81 | 66
Asthenia (General disorders) | 25 | 27
Catheter Site Pain (General disorders) | 14 | 6
Chest Pain (General disorders) | 19 | 9
Chills (General disorders) | 28 | 22
Fatigue (General disorders) | 201 | 175
Mucosal Inflammation (General disorders) | 38 | 25
Oedema Peripheral (General disorders) | 41 | 46
Pain (General disorders) | 26 | 28
Pyrexia (General disorders) | 41 | 37
Drug Hypersensitivity (Immune system disorders) | 26 | 15
Hypersensitivity (Immune system disorders) | 16 | 12
Nasopharyngitis (Infections and infestations) | 21 | 17
Sinusitis (Infections and infestations) | 38 | 21
Upper Respiratory Tract Infection (Infections and infestations) | 42 | 28
Urinary Tract Infection (Infections and infestations) | 37 | 39
Contusion (Injury, poisoning and procedural complications) | 43 | 21
Alanine Aminotransferase Increased (Investigations) | 14 | 19
Aspartate Aminotransferase Increased (Investigations) | 12 | 17
Haemoglobin Decreased (Investigations) | 30 | 21
Neutrophil Count Decreased (Investigations) | 29 | 23
Platelet Count Decreased (Investigations) | 22 | 24
White Blood Cell Count Decreased (Investigations) | 13 | 19
Decreased Appetite (Metabolism and nutrition disorders) | 48 | 61
Dehydration (Metabolism and nutrition disorders) | 18 | 13
Hyperglycaemia (Metabolism and nutrition disorders) | 23 | 17
Hypokalaemia (Metabolism and nutrition disorders) | 24 | 26
Hypomagnesaemia (Metabolism and nutrition disorders) | 39 | 35
Arthralgia (Musculoskeletal and connective tissue disorders) | 69 | 44
Back Pain (Musculoskeletal and connective tissue disorders) | 51 | 32
Bone Pain (Musculoskeletal and connective tissue disorders) | 29 | 25
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 21 | 14
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 9 | 12
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 22 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 42 | 33
Neck Pain (Musculoskeletal and connective tissue disorders) | 15 | 14
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 40 | 35
Dizziness (Nervous system disorders) | 58 | 38
Dysgeusia (Nervous system disorders) | 31 | 32
Headache (Nervous system disorders) | 119 | 70
Neuropathy Peripheral (Nervous system disorders) | 45 | 48
Peripheral Sensory Neuropathy (Nervous system disorders) | 13 | 18
Anxiety (Psychiatric disorders) | 33 | 18
Depression (Psychiatric disorders) | 37 | 24
Insomnia (Psychiatric disorders) | 51 | 36
Dysuria (Renal and urinary disorders) | 13 | 15
Proteinuria (Renal and urinary disorders) | 52 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 66 | 43
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 34 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 74 | 53
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 22 | 21
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 130 | 32
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 20 | 18
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 40 | 23
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 26 | 9
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 19 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 64 | 64
Erythema (Skin and subcutaneous tissue disorders) | 14 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 35 | 28
Rash (Skin and subcutaneous tissue disorders) | 53 | 51
Flushing (Vascular disorders) | 15 | 9
Hot Flush (Vascular disorders) | 19 | 13
Hypertension (Vascular disorders) | 102 | 20
Oral Pain (Gastrointestinal disorders) | 13 | 3
Blood Creatinine Increased (Investigations) | 13 | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 13 | 8
Hypoaesthesia (Nervous system disorders) | 9 | 12
Dry Skin (Skin and subcutaneous tissue disorders) | 13 | 6
Petechiae (Skin and subcutaneous tissue disorders) | 13 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.